CLINICAL TRIAL: NCT02948192
Title: The Reproductive Microbiome & Perinatal Health Outcome
Brief Title: The Reproductive Microbiome & Perinatal Health Outcomes
Status: Terminated | Type: Observational
Why Stopped: Inability to obtain final specimen routinely
Sponsor: Baylor Research Institute (Other)
Collaborators: Discovery Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 016-194
Record Dates: First submitted 2016-10-26; First posted 2016-10-28 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Human Microbiota; PreTerm Birth; Human Gastrointestinal Microbiota; Metabolomics
Keywords: Preterm Delivery; Preterm Birth; Vaginal Microbiome; Microbiome; Gut Microbiome; African American; Metabolomics; Pregnancy
MeSH Terms: conditions — Premature Birth | interventions — Surveys and Questionnaires; Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sample collection for bacterial microbiome identification and metabolic products
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Preterm Delivery: African american women who present for prenatal care who experience spontaneous preterm birth
  Interventions: Other: Survey, Sample collection
- Term delivery: African american women who present for prenatal care who experience term birth
  Interventions: Other: Survey, Sample collection

INTERVENTIONS:
Other: Survey, Sample collection — Survey is collected on the dietary intake of both cohorts. Sample collection is done from patients in both cohorts at multiple time points.

SUMMARY:
Pregnant African American women between 18 and 45 years of age will be enrolled at 20 weeks of gestation or less. Biological specimens (vaginal swabs, rectal swab) will be collected at enrollment, 23-24 weeks, at 28-29 weeks, and at the onset of labor. A urine sample will be obtained at entry and at the time of delivery for metabolomic analysis. Participants will also collect a dietary survey at entry, 23-24 weeks, and 28-29 weeks. The biological specimens will then be analyzed for their microbiomial profile. This will then be correlated with the timing of their delivery as well as other comorbidities such as obesity, hypertension, and diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and understand English, full decision making capabilities, African American (self-identified), Pregnant, At 20 weeks or less of gestation, Singleton pregnancy, 18-45 years of age

Exclusion Criteria:

* Race other than African American, Advanced gestational age (>20 weeks), Multiple gestations, Less than 18 years or greater than 45 years of age.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: African american women between 18 and 45 years of age who are pregnant with a singleton and present for prenatal care at 20 weeks of gestation or less.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Preterm Delivery | 36 weeks
  Onset of preterm labor with subsequent spontaneous preterm birth

SECONDARY OUTCOMES:
Microbiome profile | 36 weeks
  Evaluation of characteristics of the vaginal microbiome in cohorts
Metabolomic profile | 36 weeks
  Evaluation of characteristics of the metabolomic products present in cohort
Medical comorbidities | 36 weeks
  Evaluation of the comorbidities present in the cohort
Gut Microbiome profile | 36 weeks
  Evaluation of the characteristics of the gastrointestinal microbiome in cohorts
Term delivery | 36 weeks
  Delivery at term

IPD SHARING:
Plan to Share IPD: No